CLINICAL TRIAL: NCT05488613
Title: Healthcare Resource Utilization in Adults Diagnosed With Acute Myeloid Leukemia (AML) With a Focus on Patients Treated With Rydapt (Midostaurin) in Helsinki and Uusimaa Hospital District
Brief Title: Healthcare Resource Utilization in Adults Diagnosed With Acute Myeloid Leukemia (AML)
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CPKC412AFI02
Record Dates: First submitted 2022-08-03; First posted 2022-08-04 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute myeloid leukemia,; midostaurin,; healthcare resource utilization
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — midostaurin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Midostaurin: Midostaurin was administered in two different dosing options. Either as 2x25mg daily or 2x50mg daily.
  Interventions: Drug: Midostaurin

INTERVENTIONS:
Drug: Midostaurin — Midostaurin was administered in two different dosing options. Either as 2x25mg daily or 2x50mg daily.
  Other Names: Rydapt

SUMMARY:
This was a non-interventional, retrospective registry study, utilizing electronic health record (EHR) data collected in the hospital district of Helsinki and Uusimaa (HUS). Real-world health care resource utilization (HCRU) of AML patients was characterized.

DETAILED DESCRIPTION:
Adult patients (18 years or older) with the inclusion diagnosis, AML (ICD-10 C92.0), between 1.1.2013 - 30.6.2020 were followed from the index date (first ever record of the inclusion diagnosis) until the end of follow-up (30.6.2020), or death. This study did not involve any contacts to patients.

The study inclusion period was changed from 1.1.2013 - 30.6.2020 specified in the protocol to 1.1.2016 - 30.6.2020 due to lack of medication data from pre-2016.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with acute myeloid leukemia (ICD-10 C92.0) during 1.1.2016-30.6.2020
* Adult (18 years or older) at the time of first diagnosis
* Health registry data is available and accessible
* Resident in the hospital district HUS at the time of index diagnosis

Exclusion Criteria:

- AML patients with no treatment information

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (18 years or older) with Acute Myeloid Lukemia
Sampling Method: Non-Probability Sample
Enrollment: 81 (Actual)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2021-01-26 (Actual)

PRIMARY OUTCOMES:
Number of patients initiating midostaurin treatment | throughout the study, approximately 5 years
  Number of patients initiating midostaurin treatment were reported.

SECONDARY OUTCOMES:
Number of patients who received Midostaurin at induction and consolidation phases | throughout the study, approximately 5 years
  Number of patients who received Midostaurin at induction and consolidation phases were reported.
Duration of Midostaurin at induction and consolidation phase | throughout the study, approximately 5 years
  Duration of Midostaurin at induction and consolidation phase were reported.
Median average dose intensity in midostaurin treatment in induction and consolidation phase | throughout the study, approximately 5 years
  Median average dose intensity in midostaurin treatment were reported.
Most frequent comorbidities at the time of AML diagnosis | throughout the study, approximately 5 years
  Most frequent comorbidities at the time of AML diagnosis were reported.
Number of patients at the time of diagnosis (All treated AML patients) | throughout the study, approximately 5 years
  Number of patients at the time of diagnosis (All treated AML patients) were reported.
Number of AML patients receiving midostaurin consolidation treatment in inpatient or outpatient care (based on given prescriptions) | throughout the study, approximately 5 years
  Number of AML patients receiving midostaurin consolidation treatment in inpatient or outpatient care (based on given prescriptions) were reported.
Mean HCRU and related costs in different disease stages | throughout the study, approximately 5 years
  Estimate HCRU and related costs in different disease stages were reported.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for CPKC412AFI02 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17967